CLINICAL TRIAL: NCT06708390
Title: Single-Incision Laparoscopic Cholecystectomy with Inflexible Laparoscopic Instruments and Laparoscopy: a Single-Center Experience
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1092
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Benign Gallbladder Disease
Keywords: single-incision laparoscopic; laparoscopic cholecystectomy; cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SILC: single-incision laparoscopic cholecystectomy
- CLC: conventional laparoscopic cholecystectomy

SUMMARY:
Since being introduced by Mühe in 1985, laparoscopic cholecystectomy (LC) has garnered global acceptance and defined as gold standard treatment for benign gallbladder diseases (BGDs). Minimally invasive surgery technique was applied in a spectrum of surgeries including LC, namely single-incision laparoscopic cholecystectomy (SILC), initially reported by Navarra in 1997. By then this technique developed dramatically in aspects of both operation and instruments. Previous experiences with SILC across various centers have consistently demonstrated its robust safety and feasibility. Numerous clinical trials have highlighted the benefits of SILC over conventional laparoscopic cholecystectomy (CLC), particularly in terms of promoted aesthetic outcomes, reduced postoperative pain, and shorter hospital stays.However, discrepancies in postoperative complications including incisional hernias have sparked debate regarding the merits and drawbacks of SILC. Consequently, further research is urgent with larger cohorts and extended postoperative follow-up periods for a definitive assessment of SILC.

In the present study LC was performed in cases from January 2023 to March 2024, aiming to compare the overall outcomes and complications between CLC and SILC. All surgical instruments and laparoscopy were introduced through a single intraumbilical incision in SILC group, allowing the resultant scar to be discreetly concealed within the reconstructed navel. Furthermore, historical implementations of SILC have predominantly utilized specialized and novel instruments. This reliance on special equipment limited the technique's applicability and benefits in settings with more rudimentary clinical facilities. The authors successfully applied conventional laparoscopic instruments and a 10mm laparoscopy with straight and inflexible properties and simplified the surgical process. Moreover, the single-incision port used were made on site from basic stuffs and materials easily obtained from operation room.

ELIGIBILITY:
Inclusion Criteria:

* Gallbladder stone；
* Acute cholecystitis；
* Chronic cholecystitis；
* Gallbladder adenomyomatosis；
* Gallbladder polyp.

Exclusion Criteria:

* Combined with liver cirrhosis (Child grade B and above)；
* Gallbladder gangrene perforation;
* Changes in surgical plan (conversion to laparotomy,cholangiography, bile duct exploration, bile duct injury repair, abscess clearance, multivisceral resection.);
* patients and their families do not agree with the treatment lost follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with benign gallbladder diseases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | Six months postoperatively
  Postoperative complications were graded using Clavien-Dindo classification system
  .

SECONDARY OUTCOMES:
Postoperative quality of life | Six months postoperatively
  The quality of life of patients after operation was evaluated according to SF-36 。Scores in 0 to 100, the higher the score, the higher the quality of life.
Scar assessment | One month postoperatively
  Scar assessment was conducted postoperatively using Vancouver Scar Scale.The highest score was 18 points, and the lowest score was 0 points. The higher the score, the more serious the scar condition, and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Daren Liu, MD, PhD, Study Director — Chief Physician
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No